CLINICAL TRIAL: NCT07068009
Title: Testing the Training Programme on Data-driven Quality Development for Swiss Long-Term Care Facilities: A Pilot Study Within the National Implementation Programme NIP-Q-UPGRADE
Brief Title: Training and Support Programme on Data-driven Quality Development for Swiss Long-Term Care Facilities (NIP-Q-UPGRADE Subaim 2.6)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Collaborators: University of Basel (Other); University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Nathalie Wellens, Prof. Dr. Nathalie I.H. Wellens, Institut et Haute Ecole de la Santé la Source
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NIP-Q-UPGRADE WP 2.6
Record Dates: First submitted 2025-04-10; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Training; Quality of Care; Quality Indicators, Health Care; Long Term Care; Pain Assessment; Malnutrition in Elderly; Weight Loss; Physical Restraints; Benchmark
Keywords: quality indicators; long-term care; data-driven quality development; implementation; NIP-Q-UPGRADE; aged; leadership training; pilot study; benchmark
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: The study addresses long-term care facilities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training and Support Program on Data-driven Quality Development (Experimental): All participating facilities will be offered the same training and support program
  Interventions: Behavioral: Training and Support Programme on Data-driven Quality Development

INTERVENTIONS:
Behavioral: Training and Support Programme on Data-driven Quality Development — The training and support program uses a train-the-trainer strategy.
  The research team:
  * develop training and support materials
  * organize an e-mail helpdesk support
  * organize and conduct the scientific examination
  The external training providers:
  - train the management representatives and the quality leaders.
  The quality leader and the manager:
  * elaborate and test a quality development project based on one MQI with PDCA cycle
  * animate interprofessional meetings
  * organize a collective workshop with residents and relatives
  * engage residents and relatives in individual conversations by testing a brochure

SUMMARY:
Since 2019, long-term care facilities (LTCFs) in Switzerland have been required by the Federal Insurance Law (KVG, Art. 59a) to report data for the calculation and public reporting of medical quality indicators (MQIs) in four clinical domains: polypharmacy, pain, malnutrition, and physical restraints. This data serves both for monitoring care quality at the national level through public reporting and for internal quality development. Contextual analysis showed that various quality development methods are already known and used in Swiss LTCFs. However, significant challenges remain: limited resources, time constraints, and restricted access to MQI data hinder effective use. Facilities reported a greater need for support in using MQI data. They also expressed interest in peer networking, structured support for applying quality methods (such as Plan Do Check Act cycles (PDCA)), and practical tools such as training, best-practice examples, and additional resources. Residents and relatives also expressed a strong interest in being more involved in decision-making and care quality discussions.

The overall aim of the current study is to test a quality development training programme that supports LTCFs in using MQI data for continuous data-driven care quality development.

The study is structured into three thematic areas:

1. MQI Results Literacy - Supporting LTCFs in interpreting MQI reports and benchmarks.
2. Impactful Actions - Supporting LTCFs to translate MQI results into concrete quality development actions using PDCA cycles.
3. Sparking Culture - Integrating data-driven quality development into everyday practice and fostering a culture of continuous development, with a strong emphasis on strengthening the involvement of residents, relatives, and leadership.

The study follows a train-the-trainer strategy. Trainers instructed by the NIP-Q-UPGRADE research team provide structured training and coaching to Quality Leaders and management representatives of LTCFs. Quality Leaders then support their co-workers in quality development. The training programme consists of online and in-person trainings, training materials, practical tools, a website, guided tasks for facilities, and an email helpdesk for ongoing support.

Study outcomes: This sub-study of the NIP-Q-UPGRADE programme aims to assess the acceptability, feasibility, fidelity, and costs related to the training programme, both at the facility level and at the trainer level.

DETAILED DESCRIPTION:
A one-group experimental study is performed including a multiple methods evaluation.

Participants were recruited at two levels:

* the trainers responsible for delivering the training to the Quality Leaders and the Managers from the long-term care facilities,
* LTCF who test the training programme, select the Quality Leaders and Managers to participate in the training and who will elaborate and test a data-driven quality development project based on one MQI with the PDCA cycle within their facility.

The external training providers have experience in training staff in long-term care facilities. They have been instructed by the research team (February 2025) on how to conduct the developed training for facility Quality Leaders and managers. The trainings are conducted in three languages all regions of Switzerland. The research team informs the training participants about the study and the data collection.

At facility level, six to twelve LTCFs per Swiss language region (German, French and Italian speaking) were recruited between November and December 2024 (25 facilities in total over all language regions). At least two persons per facility will be trained between March and June 2025 to act as a Quality Leader or a Manager and perform tasks (1 full day in-person training and one peer-to-peer online meeting (2h) for managers; 2 full day in-person training onsite, two online workshops (3-4h), and two peer-to-peer online meetings (2x2h) for quality leaders.

In LTCFs the investigators aim to collect data from the quality leaders, the managers, the direct care staff, the broader staff and the residents and relatives. All individual participants will be asked written consent for data collection. This study examines the tested "training and support programme" during a 3-months interval, from end of March until June 2025. Data will be collected between March 2025 and August 2025.

At the training provider level

Quantitative data:

Activity logs: The costs of organizing and delivering the trainings will be assessed by using activity logbooks filled in continuously by the staff organizing and conducting the training (March to June 2025)

Qualitative data:

Group discussion: Acceptability, feasibility, fidelity, and adaptations to the training and support material, and barriers and facilitators to the implementation of the training will be assessed through group discussions with the staff involved after each of the training sessions (March to June 2025, in total 21 interviews or group discussions, 7 per language region).

At the long-term care facility level Staff level

Quantitative data:

Online survey: Acceptability, feasibility and fidelity will be assessed via surveys of involved staff at different levels in March 2025 (quality leaders and managers) and in June 2025 (quality leaders, managers, care staff and broader staff). The surveys will also ask for background information on the facilities and participants. Survey data will be collected in a secure online electronic data collection platform (REDCap).

Activity logbooks: Costs associated with the implementation will be assessed by using activity logbooks filled in by the quality leaders and managers and salary categories.

Qualitative data:

Focus groups: Acceptability, feasibility, fidelity, and adaptations to the toolkit, and barriers and facilitators to implementation will be assessed through focus group per language region per staff group mixing facilities:

1. 1 focus groups with quality leaders (June 2025, 1 per language region)
2. 1 focus groups with nurses and care staff exposed to the training and support program (June 2025, 1 per language region) Residents and relatives' level

Qualitative data:

Focus groups or interviews: Experiences, perceptions, expectations regarding their involvement in quality development during the pilot.

ELIGIBILITY:
Inclusion criteria:

1. Trainers:

   1. with competence in training staff of LTCFs
   2. with knowledge. on the current MQIs and PDCA cycle.
2. Long-term care facilities:

   1. with a cantonal recognition as a residential long-term care facility
   2. willing to implement the training and support program
   3. which can nominate at least one quality leader and one management representative
3. Quality leaders:

   1. Long-term care facility employees motivated to take up the role
   2. having sufficient knowledge of the residents, infrastructure and care processes in the facility.
   3. Ideally with experience in leadership, coordination, experience in care, datas, e.g., nurse, nurse expert, quality manager, clinical nurse specialist.
4. Management representative:

   1. any level of management staff in long-term care facility e.g., Members of the direction, health, director, nursing managers, ward leaders, facility or department managers.
   2. directly involved in supporting the implementation of the toolkit or exposed to its content
5. Nursing and care staff:

   1. Any level of nursing or care staff e.g., registered nurses, licensed practical nurses, nurse aids, care and community health assistant, providing direct care on all the MQI themes and are in direct dialogue with residents and relatives
   2. exposed to the content of the toolkit (i.e., participation in an interprofessional meeting, as a key person to co-elaborate the quality development project, participating in the testing phase of the quality development project).
6. Broader staff:

   1. Any level of broader staff e.g., non-clinical staff (e.g. sociocultural, catering, hotel service, occupational therapist, chaplaincy, stewardship, administration, technical department, dietician, medical doctors, socio-cultural team, ...), who are involved in quality goals.
   2. exposed to the content of the toolkit (i.e., participation in an interprofessional meeting, as a key person to co-elaborate the quality development project, participating in the testing phase of the quality development project).
7. Residents and relatives:

   1. All residents and relatives of the participating facilities who are exposed to the content of the toolkit (i.e., brochure, participating in the workshop for residents and relatives).

Exclusion criteria:

1. LTCFs that are participants of the study "Data Quality and National Quality Indicators in Long-term Care Facilities: a Validation Study and Evaluation Study"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the training and support program - Survey | LTCF QUALITY LEADERS, MANAGEMENT, CARE AND BROADER STAFF: Month 3-4
  Acceptability of the training and support components will be assessed in a survey with Acceptability of Intervention Measure (AIM), a 4-item instrument measuring the acceptability of an intervention with a total score (4-20): higher scores mean a better acceptability; through a survey targeting quality leaders, managers, care staff, and broader facility staff in participating facilities.
Acceptability of the training and support program - qualitative semi-structured interviews with managers | LTCF MANAGEMENT: Month 3-4
  Acceptability of the training and support components will be assessed in qualitative semi-structured interviews with managers.
Acceptability of the training and support program - focus groups | LTCF QUALITY LEADERS & CARE STAFF: Month 3-4
  Acceptability of the training and support components will be assessed in focus groups with quality leaders and care staff.
Acceptability of the training and support program - qualitative semi-structured interviews with trainers | Week 1, 2, 4, 6, 8-10, 12-13 (After each training unit)
  Acceptability of the training and support components will be assessed in semi-structured qualitative interviews with trainers after each training unit.
Feasibility of the training and support program - Survey | LTCF QUALITY LEADERS, MANAGEMENT, CARE AND BROADER STAFF: Month 3-4
  Feasibility of training and support components will be assessed in a survey with Feasibility of Intervention Measure (FIM), a 4-item instrument measuring the feasibility of an intervention with a total score (4-20): higher scores mean a better feasibility ; through a survey targeting quality leaders, managers, care staff, and broader facility staff.
Feasibility of the training and support program - qualitative semi-structured interviews with managers | LTCF MANAGEMENT: Month 3-4
  Feasibility of the training and support components will be assessed in qualitative semi-structured interviews with managers.
Feasibility of the training and support program - focus groups | LTCF QUALITY LEADERS & CARE STAFF: Month 3-4
  Feasibility of the training and support components will be assessed in focus groups with quality leaders and care staff.
Feasibility of the training and support program - qualitative semi-structured interviews with trainers | Week 1, 2, 4, 6, 8-10, 12-13 (After each training unit)
  Feasibility of the training and support components will be assessed in qualitative semi-structured interviews with trainers after each training unit.
Implementation fidelity - survey | LTCF QUALITY LEADERS, MANAGEMENT, CARE AND BROADER STAFF: Month 3-4
  Degree of fidelity to each component (yes, partial, no) will be measured using a survey targeting quality leaders, managers, care staff, and broader facility staff.
Implementation fidelity - qualitative interviews semi-structured with managers | LTCF MANAGEMENT: Month 3-4
  Implementation fidelity of the training and support components will be assessed in qualitative semi-structured interviews with managers.
Implementation fidelity - focus groups | LTCF QUALITY LEADERS & CARE STAFF: Month 3-4
  Implementation fidelity of the training and support components will be assessed in focus groups with quality leaders and care staff.
Implementation fidelity - qualitative semi-structured interviews with trainers | Week 1, 2, 4, 6, 8-10, 12-13 (After each training unit)
  Implementation fidelity of the training and support components will be assessed in qualitative semi-structured interviews with trainers after each training unit.
Barriers to the implementation of the toolbox - focus groups | LTCF QUALITY LEADERS & CARE STAFF: Month 3-4
  Barriers to the implementation will be explored in focus groups with quality leaders and care staff, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Barriers to the implementation of the toolbox - qualitative semi-structured interviews | LTCF MANAGEMENT: Month 3-4
  Barriers to the implementation will be explored in qualitativ semi-structured interviews with managers, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Barriers to the implementation of the toolbox - qualitative semi-structured interviews with trainers | Week 1, 2, 4, 6, 8-10, 12-13 (After each training unit)
  Barriers to the implementation will be explored in qualitativ semi-structured interviews with trainers after each training unit, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Facilitators to the implementation of the toolbox - focus group | LTCF QUALITY LEADERS & CARE STAFF: Month 3-4
  Facilitators to the implementation will be explored in focus groups with quality leaders and care staff, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Facilitators to the implementation of the toolbox - qualitative semi-structured interviews | LTCF MANAGEMENT: Month 3-4
  Facilitators to the implementation will be explored in qualitative semi-structured interviews with managers, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Facilitators to the implementation of the toolbox - qualitative semi-structured interviews with trainers | Week 1, 2, 4, 6, 8-10, 12-13 (After each training unit)
  Facilitators to the implementation will be explored in qualitative semi-structured interviews with trainers after each training unit, and categorized according to the Consolidated Framework of Implementation Research (CFIR).
Sum of costs associated with implementation of the toolkit in Swiss francs | Monthly up to 3 months
  Costs will be calculated based on time spent on implementation activities per staff group with corresponding hourly salary estimate, recorded in an activity logbook

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie I.H. Wellens, Prof. Dr., Principal Investigator — Institute and School of Nursing La Source, HES-SO University of Applied Sciences Western Switzerland; Franziska Zúñiga, Prof.Dr., Principal Investigator — University of Basel
Locations (3):
- Switzerland (3):
  - Institut für Pflegewissenschaft - Nursing Science (INS), University of Basel, Basel, Basel
  - Institute and School of Nursing La Source, HES-SO University of Applied Sciences Western Switzerland, Lausanne, Canton of Vaud
  - Department of Business Economics, Health and Social Care, University of Applied Sciences and Arts of Southern Switzerland (SUPSI), Manno, Canton Ticino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.curaviva.ch/nip-q-upgrade-fr?lang=fr&redirect_lang
- See also: Related Info — https://www.ecolelasource.ch/nip-q-upgrade/